CLINICAL TRIAL: NCT03424122
Title: A Phase 1, Open-Label, Dose-Finding Study of INCB050465 in Combination With Investigator Choice of Rituximab, Bendamustine and Rituximab, or Ibrutinib in Participants With Previously Treated B-Cell Lymphoma (CITADEL-112)
Brief Title: INCB050465 in Combination With Rituximab, Bendamustine and Rituximab, or Ibrutinib in Participants With Previously Treated B-Cell Lymphoma (CITADEL-112)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-112 (CITADEL-112); Parsaclisib (Other: Incyte Corporation); 2017-004088-11 (EudraCT Number)
Record Dates: First submitted 2018-01-25; First posted 2018-02-06 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: B-cell Lymphoma
Keywords: Diffuse large B-cell lymphoma (DLBCL); follicular lymphoma (FL); marginal zone lymphoma (MZL); mantle cell lymphoma (MCL); phosphatidylinositol 3-kinase delta (PI3Kδ) inhibitor
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell | interventions — parsaclisib; Rituximab; Bendamustine Hydrochloride; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): Parsaclisib + Rituximab
  Interventions: Drug: Parsaclisib; Drug: Rituximab
- Treatment B (Experimental): Parsaclisib + Bendamustine + Rituximab
  Interventions: Drug: Parsaclisib; Drug: Rituximab; Drug: Bendamustine
- Treatment C (Experimental): Parsaclisib + Ibrutinib
  Interventions: Drug: Parsaclisib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Parsaclisib — Parsaclisib administered orally once daily for 8 weeks followed by once weekly.
  Other Names: INCB050465
Drug: Rituximab — Rituximab administered intravenously at the protocol-defined dose regimen according to treatment group.
  Other Names: Rituxan
  Arms: Treatment A; Treatment B
Drug: Bendamustine — Bendamustine administered intravenously on Days 1 and 2 of each cycle for up to 6 cycles.
  Other Names: Treanda, Bendeka
  Arms: Treatment B
Drug: Ibrutinib — Ibrutinib administered orally once daily.
  Other Names: Imbruvica
  Arms: Treatment C

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of parsaclisib when combined with rituximab, bendamustine and rituximab, or ibrutinib in participants with relapsed or refractory B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 years or older on the day of signing the Informed Consent Form (ICF).
* Histologically confirmed indolent/aggressive DLBCL, FL, MZL, or MCL.
* Participants with DLBCL, MZL or MCL must have received at least 1 prior line of systemic therapy with documented progression or documented failure to achieve CR or PR after the most recent systemic treatment regimen.
* Participants with FL must have received at least 2 prior lines of systemic therapy with documented progression or documented failure to achieve CR or PR after the most recent systemic treatment regimen.
* Ineligible for stem cell transplant.
* Participants with DLBCL must have failed or refused stem cell transplantation or failed first-line salvage therapy if ineligible for transplantation.
* Must be willing to undergo an incisional or excisional lymph node or tissue biopsy or to provide a lymph node or tissue biopsy from the most recent available archival tissue.
* Life expectancy of > 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2 (see Appendix D).
* Willingness to avoid pregnancy or fathering a child.
* Ability to comprehend and willingness to sign an ICF

Exclusion Criteria:

* Evidence of transformed non-Hodgkin lymphoma histologies (with the exception of FL).
* Histologically confirmed rare non-Hodgkin B-cell subtypes.
* History of or central nervous system lymphoma (either primary or metastatic) or leptomeningeal disease.
* Prior treatment with idelalisib, other selective PI3Kδ inhibitors, or a pan-PI3K inhibitor.
* For participants to be treated with bendamustine (Treatment B), prior treatment with bendamustine (within 12 months of the start of study treatment). Participants with prior bendamustine treatment (> 12 months before the start of study treatment) are eligible if they meet the following criteria:

  * Did not discontinue because of tolerability concerns.
  * Achieved either partial response (PR) or complete response (CR) to the bendamustine regimen of at least 12 months in duration before relapse/progression.
  * Experienced progression following a regimen containing an alkylating agent.
* For participants to be treated with ibrutinib (Treatment C), prior treatment with a Bruton's tyrosine kinase (BTK) inhibitor.
* Allogeneic stem cell transplant within the last 6 months or autologous stem cell transplant within the last 3 months before the date of the first dose of study treatment.
* Active graft-versus-host disease following allogeneic transplant.
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) | Up to approximately 12 months.
  A TEAE is any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study treatment.

SECONDARY OUTCOMES:
Apparent clearance of parsaclisibin combination with rituximab, bendamustine and rituximab, or ibrutinib | Up to approximately 1 month.
  Measured to assess the plasma pharmacokinetic profile of parsaclisib in combination with rituximab, bendamustine and rituximab, and ibrutinib.
Apparent volume of distribution of parsaclisib in combination with rituximab, bendamustine and rituximab, or ibrutinib | Up to approximately 1 month.
  Measured to assess the plasma pharmacokinetic profile of parsaclisib in combination with rituximab, bendamustine and rituximab, and ibrutinib.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, MD, Study Director — Incyte Corporation
Locations (21):
- United States (9):
  - University of Arizona Cancer Center - Out Pt., Tucson, Arizona
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Texas Oncology, Austin, Texas
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Smith Clinic, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology San Antonio, San Antonio, Texas
- Italy (4):
  - Asst Spedali Civili Di Brescia, Brescia
  - Azienda Ospedaliera San Gerardo Di Monza, Monza
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Ospedale Delle Croci - Ematologia Ravenna, Ravenna
- Spain (8):
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital General Universitari Vall D Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Hospital Universitario Hm Sanchinarro, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario Y Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No